CLINICAL TRIAL: NCT00700622
Title: A Phase3, Multi-Center, Open-Label, Randomized, Clinical Trial Evaluating the Efficacy and Safety of Technosphere® Insulin Inhalation Powder in Combination With Lantus® Versus Humalog® in Combination With Lantus® in Subjects With Type 1 Diabetes Mellitus Over a 16-Week Treatment Period
Brief Title: Safety and Efficacy of Technosphere® Insulin Inhalation Powder and Lantus® Compared to Humalog® and Lantus® Over 16-Weeks
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor stopped development of the MedTone inhaler in favor of an improved device (Gen2 inhaler)
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-117
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TI + Insulin glargine (Experimental): Technosphere Insulin Inhalation Powder in combination with Lantus (insulin glargine)
  Interventions: Drug: Technosphere Insulin
- Insulin lispro + Insulin glargine (Experimental): Humalog (insulin lispro) in combination with Lantus (insulin glargine)
  Interventions: Drug: Insulin glargine; Drug: Insulin lispro

INTERVENTIONS:
Drug: Technosphere Insulin — Technosphere Insulin Inhalation Powder 15U or 30U
  Arms: TI + Insulin glargine
Drug: Insulin glargine — Lantus-injectible supplied as 3mL (300 units) pens
  Arms: Insulin lispro + Insulin glargine
Drug: Insulin lispro — Humalog autopen cartridges pre-filled with 3mL (300 units)
  Arms: Insulin lispro + Insulin glargine

SUMMARY:
The objective of this study is to demonstrate that TI® Inhalation Powder combined with Lantus® is as effective as Humalog® combined with Lantus® on HbA1c.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 and ≤ 80 years old
* Clinical diagnosis of type 1 diabetes mellitus for more than 12 months
* Body mass index (BMI) ≤ 30 kg/m2
* Stable antidiabetic regimen of sc insulin therapy at a total daily dose ≤ 1.5 IU/kg/day
* HbA1c > 7.0% and ≤ 9.0%
* C-peptide level ≤ 0.30 pmol/mL
* Nonsmokers (includes cigarettes, cigars, pipes, and chewing tobacco) for at least the preceding 6 months
* Negative urine cotinine defined as ≤ 100 ng/mL
* Pulmonary function tests (PFTs):

  * Forced expiratory volume in 1 second (FEV1) ≥ 70% Third National Health and Nutrition Examination Survey (NHANES III) predicted
  * FEV1 as a percentage of FEV1/forced vital capacity (FVC) ≥ 70% (NHANES III) predicted
  * Total lung capacity (TLC) ≥ 80% predicted (Intermountain Thoracic Society [ITS])
  * Single breath carbon monoxide diffusing capacity of the lung, hemoglobin-corrected (DLco-Hb) (uncorrected) ≥ 70% predicted
* For the subset of subjects having Doppler echocardiograms: right ventricular systolic pressure (RVSP) ≤ 40 mm Hg at Visit 1
* Written informed consent

Exclusion Criteria:

* Treatment with any type of antidiabetic drugs, other than sc insulin, within the preceding 12 weeks
* Two or more severe hypoglycemic episodes within 6 months of screening or episode of severe hypoglycemia between Visit 1 and Visit 5
* Any hospitalization or emergency room visit due to poor diabetic control within 6 months of Visit 1, or hospitalization or emergency room visit due to poor diabetic control between Visit 1 and Visit 5
* Severe complications of diabetes, in the opinion of the PI, including symptomatic autonomic neuropathy; disabling peripheral neuropathy; active proliferative retinopathy; nephropathy with renal failure, renal transplant, or dialysis; history of foot ulcers; nontraumatic amputations due to gangrene; or vascular claudication
* Previous exposure to an inhaled insulin product within 3 months of Visit 1
* History of insulin pump use within 6 weeks of Visit 1
* Allergy or known hypersensitivity to insulin or to any of the drugs to be used in the trial, or a history of hypersensitivity to TI Inhalation Powder or to drugs with a similar chemical structure
* Significant improvement in pre- to postbronchodilator spirometry at Visit 1 (defined as an increase of 12% and 200 mL in either FEV1 or FVC)
* History of chronic obstructive pulmonary disease (COPD), clinically proven asthma, or any other clinically important pulmonary disease (eg, obstructive sleep apnea) confirmed by pulmonary function testing or radiologic findings
* Inability to perform spirometry maneuvers meeting recommended American Thoracic Society (ATS) standards of acceptability and repeatability criteria
* Active respiratory infection (subject could return after 30 days from resolution for rescreening); if respiratory infection manifested after Visit 1 but before Visit 1 PFTs, subject was to be scheduled for PFTs after 30 days from resolution of respiratory infection. An additional hemoglobin was to be required
* Major organ system diseases, including:

  * Seizure disorder
  * Significant cardiovascular dysfunction or history within 3 months of Visit 1, eg, congestive heart failure (New York Heart Association [NYHA] Class III or IV), or serious arrhythmia, myocardial infarction, cardiac surgery, recurrent syncope, transient ischemic attacks, or cerebrovascular accident
  * Uncontrolled hypertension with a systolic blood pressure > 180 mm Hg or diastolic blood pressure > 110 mm Hg at Visit 1 despite pharmacologic treatment
  * Nephrotic syndrome; renal dysfunction or disease; serum creatinine > 2.0 mg/dL (0.11 mmol/L) in men and > 1.8 mg/dL (0.1 mmol/L) in women; or blood urea nitrogen (BUN) > 50 mg/dL (2.8 mmol/L)
  * Cancer (other than excised cutaneous basal cell carcinoma) within the past 5 years or any history of lung neoplasms
  * History of active viral or cirrhotic hepatic disease or abnormal liver enzymes as evidenced by serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 3 times the upper limit of normal (ULN)
  * Active infection (eg, human immunodeficiency virus [HIV], hepatitis) or history of severe infection within 30 days of Visit 1
  * Anemia (hemoglobin ≤ 10.5 g/dL for women or ≤ 11.5 g/dL for men)
  * Diagnosis of systemic autoimmune or collagen vascular disease requiring previous or current treatment with systemic corticosteroids, cytotoxic drugs, or penicillamine
  * Any concurrent illness, other than diabetes mellitus, not controlled by a stable therapeutic regimen
* Current or previous chemotherapy or radiation therapy that might result in pulmonary toxicity
* Use of medications prescribed for weight loss (eg, sibutramine, orlistat) within 12 weeks of Visit 1
* Any history of or current use of amiodarone
* Clinically significant abnormalities on screening laboratory evaluation (unless discussed with and approved by the medical monitor)
* Women who were pregnant, lactating, or planning to become pregnant during the trial
* Women of childbearing potential (defined as premenopausal and not surgically sterilized or postmenopausal for fewer than 2 years) not practicing adequate birth control. Adequate birth control was defined as using oral, percutaneous, or transdermal contraceptives; condoms and diaphragms (double barrier) with a spermicide; or intrauterine devices. Postmenopausal for this trial included amenorrhea for 2 or more years or surgically sterile
* Current drug or alcohol abuse or a history of drug or alcohol abuse that, in the opinion of the PI, would make the subject an unsuitable candidate for participation in the trial
* Exposure to any investigational medications or devices within 30 days before trial entry, or participation in another clinical trial while participating in this trial
* Unable or unlikely to comprehend and follow the trial protocol (including SBGM and diabetes education)
* Unable or unlikely to comprehend how to use the MedTone Inhaler or inability to use the device
* Unable or unlikely to follow a meal plan that included at least 2 meals/day (with or without a third meal or additional snacks)
* Noncompliance with medication or procedures that, in the PI's opinion, might affect the trial data or subject safety and that precluded the subject from further participation in the trial
* Any other concurrent medical or major psychiatric condition that, in the opinion of the PI, made the subject unsuitable for the clinical trial or could limit the validity of the informed consent or impair the subject's ability to participate in the trial
* For the subset of subjects having Doppler echocardiograms:

  * Subjects with left ventricular ejection fraction (LVEF) ≤ 35% at Visit 1
  * Subjects with known history of sickle cell disease
  * Previous use of Redux® (dexfenfluramine) or Pondimin® (fenfluramine)
  * History of valvular heart disease, including mild or greater aortic insufficiency or moderate or greater mitral insufficiency
  * Significant cardiovascular dysfunction or history within 12 months of Visit 1 (eg, congestive heart failure [NYHA Class III or IV]) or serious arrhythmia, treatment with medications to control or treat arrhythmias, myocardial infarction, cardiac surgery, recurrent syncope, transient ischemic attacks, or cerebrovascular accident
  * History of pulmonary embolism or deep venous thrombosis in the 12 months before Screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-05; Primary Completion 2009-11 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (20):
  - Diabetes/Lipid Management and Research Center, Huntington Beach, California
  - The Whittier Institute for Diabetes Clinical Trials, La Jolla, California
  - Dorothy L & James E Frank Diabetes Research Institute, San Mateo, California
  - Barbara Davis Center for Diabetes Young Adult Clinic, Aurora, Colorado
  - University of Miami Diabetes Research Institute, Miami, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Washington University School of Medicine, St Louis, Missouri
  - Deaconess Billings Clinic Research Center, Billings, Montana
  - Mountain Diabetes & Endocrine Center, Asheville, North Carolina
  - Endocrine Research Physicians East PA, Greenville, North Carolina
  - Your Diabetes Endocrine Nutrition Group, Inc., Mentor, Ohio
  - OHSU Diabetes Center Research Oregon Health & Science University, Portland, Oregon
  - AM Diabetes and Endocrinology Center, Barrtlett, Tennessee
  - Dallas Diabetes & Endocrine Center, Dallas, Texas
  - Baylor Endocrine Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Diabetes Research Center -Fletcher Allen Health Care, South Burlington, Vermont
  - Diabetes Care Center, Seattle, Washington
- Brazil (2):
  - Centro de Pesquisas em Diabetes Ltda, Porto Alegre, Rio Grande do Sul
  - CPClin-Centro de Pesquisas Clinicas, São Paulo, São Paulo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The FPFV was May 30, 2008. Multinational trial conducted in the US and Brazil.
Pre-assignment Details: 2 week screening period prior to randomization - 276 Screened / 138 Eligible. 130 subjects were randomized; 138 screen failures and 8 discontinued prior to randomization.
Period: Overall Study
Arm/Group | TI + Insulin Glargine | Insulin Lispro + Insulin Glargine
Started | 65 | 65
Completed | 52 | 60
Not Completed | 13 | 5
Not completed — Adverse Event | 4 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Other | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TI + Insulin Glargine | Insulin Lispro + Insulin Glargine | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (11.82) | 39.4 (11.46) | 39.0 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 32 | 57
  Male | 40 | 33 | 73
Weight [Mean (Standard Deviation); unit: kg] | 74.49 (13.270) | 74.18 (13.894) | 74.3 (13.53)
Height [Mean (Standard Deviation); unit: cm] | 172.22 (9.238) | 169.61 (9.807) | 170.9 (9.579)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.07 (3.744) | 25.63 (3.141) | 25.3 (3.454)
HbA1c [Mean (Standard Deviation); unit: %] | 7.76 (0.550) | 7.62 (0.602) | 7.69 (0.579)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 86.26 (10.445) | 87.31 (10.669) | 86.78 (10.530)
Fasting Blood Glucose [Mean (Standard Deviation); unit: mg/dL] | 178.06 (76.916) | 176.20 (67.268) | 177.15 (72.084)
Race [Number; unit: participants]
  Caucasian | 56 | 59 | 115
  Black | 3 | 0 | 3
  Hispanic | 5 | 5 | 10
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c to Week 16
Description: Change from Baseline in glycosylated hemoglobin at Week 16
Time Frame: Baseline to Week 16
Population: Intent to Treat with Available Data at Week 16
Measure: Least Squares Mean (Standard Error); unit: percentage of total hemoglobin
Arm/Group | TI + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 52 | 58
percentage of total hemoglobin | -0.10 (0.087) | -0.03 (0.082)
Statistical Analysis 1: Comparison: Insulin Lispro + Insulin Glargine; Test type: Non-Inferiority or Equivalence — A sample size of 92 subjects in each group was required to complete the trial. Approximately 230 subjects were to be randomized to achieve 184 completers (assuming a 20% dropout rate). This would have provided 80% power for a noninferiority design to test the difference of a 4-month change in HbA1c levels between treatment groups, assuming the upper noninferiority margins Δ of 0.5% with a standard deviation of 1.2 and a 1-sided alpha of 0.025; ANCOVA; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.31 to 0.17], Standard Error of Mean 0.119

ADVERSE EVENTS:
Time Frame: SAEs: From first dose to 30d post last dose AEs: From first dose to 30d post last dose
Arm/Group | TI + Insulin Glargine | Insulin Lispro + Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 1/65 | 3/65
Other Adverse Events (participants affected / at risk) | 42/65 | 34/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TI + Insulin Glargine (N=65) | Insulin Lispro + Insulin Glargine (N=65)
Delayed recovery from anesthesia (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 2
Hypoglycemic seizure (Metabolism and nutrition disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TI + Insulin Glargine (N=65) | Insulin Lispro + Insulin Glargine (N=65)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 0
Hypoglycaemia (Endocrine disorders) | 21 | 23
Sinusitis (Infections and infestations) | 5 | 2
Upper respiratory infection (Infections and infestations) | 5 | 6
Chest discomfort (General disorders) | 4 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Influenza (Infections and infestations) | 3 | 11
Nasopharyngitis (Infections and infestations) | 3 | 4

LIMITATIONS AND CAVEATS:
- Early termination of trial leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MannKind has right to 1st joint multicenter publication. After 1st publication PI may publish data only if PI submits proposed publication to MNKD for review 60 days prior to publication date. MNKD may remove any confidential information. If a multicenter publication is not submitted 12 months after conclusion, abandonment, or termination of the study at all sites, or if MNKD confirms there will be no multicenter Study publication, PI may publish the study results subject to MNKD rights herein.